CLINICAL TRIAL: NCT01683149
Title: Phase I, Traditional 3+3, Trial of PO Sorafenib and Topotecan in Refractory or Recurrent Pediatric Solid Malignancies
Brief Title: Sorafenib and Topotecan in Refractory/Recurrent Pediatric Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pediatric Cancer Foundation (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16963; ONC-2011-49 (Other: Bayer HealthCare); Sunshine Project 002 (Other Grant/Funding Number: Pediatric Cancer Foundation)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Solid Tumor
Keywords: Refractory; Relapsed; Recurrent; Pediatric; Malignancy
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Topotecan; Topoisomerase I Inhibitors; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Chemotherapy (Experimental): Combination Chemotherapy: Topotecan and Sorafenib. Participants will receive the treatment in cycles. Every cycle is 28 days long. For the first cycle participants will get the chemotherapy drugs:
  * Topotecan PO (by mouth) once daily on days 1-5 and days 8-12
  * Sorafenib PO (by mouth) twice daily (BID), continuously on days 2-28 of cycle one and days 1-28 on each additional cycle.
  * Level -1: Topotecan 1.0 mg/m^2: Sorafenib 100 mg/m^2 BID
  * Level -2: Topotecan 0.8 mg/m^2: Sorafenib 100 mg/m^2 BID
  * Level 1: Topotecan 1.0 mg/m^2: Sorafenib 150 mg/m^2 BID
  * Level 2: Topotecan 1.4 mg/m^2: Sorafenib 150 mg/m^2 BID
  * Level 3: Topotecan 1.4 mg/m^2: Sorafenib 200 mg/m^2 BID
  * Level 4: Topotecan 1.8 mg/m^2: Sorafenib 200 mg/m^2 BID
  Interventions: Drug: Topotecan; Drug: Sorafenib

INTERVENTIONS:
Drug: Topotecan — Topotecan will be given by mouth as outlined in treatment arm.
  Other Names: Topoisomerase-I inhibitor
Drug: Sorafenib — Sorafenib will be given by mouth as outlined in treatment arm.
  Other Names: BAY 43-9006

SUMMARY:
H. Lee Moffitt Cancer Center and Research Institute will be the Sunshine Project Coordinator, but will not be recruiting locally.

The purpose of this research study is to establish a dose of the combination of drugs, Topotecan and Sorafenib in children. This will be called the maximum tolerated dose. The chemotherapy in this study is a combination of Topotecan and Sorafenib. The investigators are trying to find the highest dose of Topotecan and Sorafenib that can be given safely to children with Refractory or Recurrent Pediatric Solid Malignancies. The investigators will do this by testing different doses of these drugs in different groups of children. The investigators will also study how the body processes these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks (3 months)
* Must have had relapsed or refractory solid tumor malignancy, or a relapsed or refractory central nervous system malignancy AND must have received at least one prior course of therapy for their malignancy.
* Patients with a solid tumor must have radiographic evidence of disease. Bone only disease is acceptable if biopsy proven but will not be eligible for response criteria by RECIST 1.1. Ideally patients will have disease evaluable by RECIST 1.1.
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Karnofsky ≥ 50 for patients > 16 years of age, and Lansky ≥ 50 for patients ≤ 16 years of age.
* Prior Therapy: Patients with solid tumors must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Previous Sorafenib or Topotecan: Patients may not have previously been treated with sorafenib. Patients may have been previously treated with topotecan provided it was in combination with other agents and the most recent dose was more than 6 months from study entry. Patients in whom disease has progressed on single agent topotecan will not be eligible for this study.
  2. Myelosuppressive Chemotherapy: Patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks or nitrosourea within 6 weeks of entry onto this study.
  3. Hematopoietic Growth Factors: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.
  4. Biologic (anti-neoplastic agent): At least 21 days or 5 half lives (whichever is greater duration) since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
  5. Radiation Therapy (XRT): ≥ 4 wks for local palliative XRT (small port); ≥ 3 months must have elapsed if prior TBI, or craniospinal XRT or if ≥ 50% radiation of pelvis; ≥ 6 weeks must have elapsed if other substantial bone marrow (BM) radiation.
  6. Stem Cell Transplant or Rescue without total body irradiation (TBI): For allograft: no evidence of active graft vs. host disease and ≥ 3 months must have elapsed since stem cell transplantation (SCT). Autologous transplant recipients must be transfusion independent and not require growth factors for >4 weeks.
* All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate will be obtained according to local Institutional Review Board (IRB) guidelines. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Organ Function Requirements - Adequate Bone Marrow Function Defined As:

  1. Peripheral absolute neutrophil count (ANC) ≥ 1500/μL.
  2. Platelet count ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
  3. Hemoglobin ≥ 10.0 gm/dL (may receive red blood cell transfusions)
  4. Patients with known bone marrow metastatic disease will be eligible for study. These patients must not be known to be refractory to red cell or platelet transfusion. If dose limiting hematologic toxicity is observed, all subsequent patients enrolled at the dose level must not have bone marrow metastatic disease.
* Adequate Renal Function Defined As: Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 60ml/min/1.73 m^2, or serum creatinine based on age/gender as defined in the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).
* Adequate Liver Function Defined As:

  1. Bilirubin (sum of conjugated + unconjugated) ≤ upper limit of normal (ULN) for age
  2. Alanine transaminase (ALT) ≤ upper limit of normal for age
  3. All clinically significant chemistries excluding alkaline phosphatase, uric acid, aspartic transaminase (AST) and lactate dehydrogenase (LDH) must be grade 1 or less
* Adequate Cardiac Function Defined As:

  1. Normal 12 lead EKG with corrected QT interval (QTc) < 450 msec, and either:
  2. Shortening fraction ≥ 28% or left ventricular ejection fraction ≥ 50%.
  3. Systolic Blood Pressure and Diastolic Blood Pressure ≤ 95th percentile for age and gender
* Adequate Pulmonary Function Defined As: No evidence of dyspnea at rest, and a resting pulse oximetry > 92%.
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of enrollment, signing the Informed Consent Form (ICF).
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Prothrombin time-international normalized ratio (PT-INR) ≤ 1.5 X ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN.
* Participants (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug.
* Must be able to swallow and retain oral medication

Exclusion Criteria:

* Previous assignment to treatment during this study
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management
* Evidence or history of bleeding diathesis or coagulopathy
* Any pulmonary hemorrhage/bleeding event of NCI-CTCAE v4.0 Grade 2 or higher within 4 weeks of treatment; any other hemorrhage/bleeding event of NCI-CTCAE v4.0 Grade 3 or higher within 4 weeks of treatment
* Have used strong cytochrome P450 3A4 (CYP3A4) inducers (eg, phenytoin, carbamazepine, phenobarbital, St. John's Wort [Hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) within 28 days before treatment
* Any previously untreated or concurrent cancer that is distinct in primary site or histology from the primary. Patients surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed. All cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form)
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* History of organ allograft. (Including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Women who are pregnant or breast-feeding
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments
* Any condition which, in the investigator's opinion, makes the patient unsuitable for trial participation

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 24 months
  Establish the recommended phase II dose of the combination of topotecan and sorafenib in children. This will be the maximum tolerated dose.

SECONDARY OUTCOMES:
Time to Progression (TTP) | 24 months
  Determine Time to Progression (TTP) for all patients, comparing TTP on study to TTP on previous regimen. This study will use the (RECIST 1.1) Response Evaluation Criteria in Solid Tumors from the NCI for assessment of radiographic response in patients with solid tumors and in order to determine if patients have met off study criteria, i.e. disease progression. Progressive Disease (PD): At least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions, or evidence of laboratory or clinical progression.
The Number of Participants with Adverse Events as a Measure of Safety and Feasibility | 24 months
  Describe the toxicity as per NCI Common Toxicity Criteria, version 4.0 (CTCAE 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Damon Reed, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; G. Douglas Letson, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (9):
- United States (9):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Connecticut Childrens Medical Center, Hartford, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Delaware, Wilmington, Delaware
  - University of Florida, Gainesville, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Jacksonville, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - All Children's Hospital, St. Petersburg, St. Petersburg, Florida
  - Montefiore Medical Center, Children's Hospital at Montefiore, The Bronx, New York
  - Primary Children's Medical Center/Utah, Salt Lake City, Utah